CLINICAL TRIAL: NCT06581458
Title: Home Transcranial Direct-Current Stimulation for Motoric Cognitive Risk Syndrome
Acronym: HometDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 0098-24-TLV
Record Dates: First submitted 2024-07-03; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Motoric Cognitive Risk Syndrome
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS immediate intervention group (Experimental): Participants in the tDCS Immediate Intervention Group will receive an initial two-week period of transcranial Direct Current Stimulation (tDCS) treatment. This will be followed by three months of continued tDCS intervention.
  Interventions: Drug: tDCS
- Late intervention group (tDCS+ sham) (Sham Comparator): Participants in the Late Intervention Group will first receive a placebo (sham) treatment for three months. This will be followed by a two-week period of active transcranial Direct Current Stimulation (tDCS) treatment, then three months of continued tDCS intervention.
  Interventions: Drug: tDCS

INTERVENTIONS:
Drug: tDCS — The immediate intervention group will continue to receive five tDCS treatments per week for 6 months. The late intervention group will receive five sham treatments per week for 3 months and then begin receiving five weekly tDCS treatments for an additional 3 months.

SUMMARY:
1. To examine the effect of a two-week tDCS intervention of 3 months of continued tDCS intervention versus 3 months of receiving a placebo treatment (dummy). On the costs of performing an action task (dual task cost) walking speed, cognitive measures and motor function.
2. To examine whether the effects of tDCS build up over time by creating a delayed start mechanism in the intervention (delayed-start design)
3. Examining mechanical and neuroplastic effects of tDCS intervention
4. To examine the response to tDCS over time

DETAILED DESCRIPTION:
* The study aims to investigate the mechanical and neuroplastic effects of a tDCS intervention.
* The intervention consists of an initial two-week period of tDCS application, followed by three months of continued tDCS treatment.
* A placebo group will receive a dummy treatment for three months to compare the outcomes.
* The study will measure various parameters including the costs of performing an action task (dual task cost), walking speed, cognitive measures, and motor function.
* A delayed-start design will be used to determine if the effects of tDCS build up over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-90
* Cognitive complaints

  * A positive answer to the question "Do you feel you have more problems than most people?"
  * A negative answer to the question "Is your thinking as clear and sharp as it was before?"
* Slow walking - one standard deviation below the average for age and gender (under age 75: men less than 101.9 cm/s, women less than 97.4 cm/s. Over or equal to age 75: men less than 85.3 s) m/s women less than 76.7 cm/s)
* No significant disability

  * There is the ability to walk without support on a walking carpet
  * A result below 9 in the Functional Activities Questionnaire index
* Identification as qualified
* Identification as willing and able to operate a tDCS device or have a partner who is able to operate the device during home use. According to the criteria:

  * Inclusion: selected by the patient, over the age of 21, with basic computer skills and available throughout the study period
  * Exclusion: MOCA score lower than or equal to 26. Presents insufficient understanding, poor vision, severe joint problems in the hands, deformity pain or other conditions that may interfere with the successful operation of the tDCS
* Has access to a reliable wireless internet network (WiFi) at the patient's home

Exclusion Criteria:

* Less than eight years of study
* dementia

  * According to the clinical definition clinical dementia rationing (CDR) score 1 or higher
  * Previous diagnosis
  * Performance in the range indicating dementia in the neuropsychological test bettery (lower than 2 standard deviations below the age- and sex-matched average)
* IQ is low or equal to 85 in the WTAR test. without a background of mental disability
* Current diagnosis of major psychiatric disorders (schizophrenia, bipolar, major depression)
* Evidence of moderate to severe symptoms of depression. A score high or equal to 9 on the 15 item geriatric depression scale
* History of head injury that led to prolonged loss of consciousness
* History of palpitations of unknown origin that may indicate convulsions
* History of convulsions, diagnosis of epilepsy in the patient or in most of the first degree family. Except for a case of a single seizure of benign etiology determined by a neurologist
* Hospitalization during the last three months following an acute illness or musculoskeletal injury with a significant impact on walking or stability
* An unbalanced medical condition that can worsen following convulsive stimulation (cardiac malformation, cardiac arrhythmias, asthma, etc.)
* Substance use disorders during the last six months
* A wig or hair design that prevents contact of the electrodes with the scalp or interferes with the administration of the stimulation
* Chronic vertigo
* A cardiac event within the last six months
* Active cancer treated with chemotherapy or radiation
* blindness
* Visual hallucinations (according to history or self-report)
* There are contraindications for MRI or tDCS as defined by the International Federation for Clinical Neurophysiology

  * Includes unprovoked convulsions during the last 2 years
  * Danger of finding ferromagnetic objects in the body, self-reporting of medical implants in the body (DBS, deep brain stimulation, drug delivery pump, cochlear implant, pacemaker)
  * Inventions active dermatological condition
* History of behavior disorders in REM sleep, sometimes an early sign of Parkinson's disease
* Medications and medical history will be examined by a clinician and a decision regarding entry into the study will be based on medical history, current medication dosage and medication change before or during the treatment as well as combination with other active CNS medications.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy in Serial Subtractions Task | 45-second
  articipants will perform serial subtractions from a random 3-digit number between 200 and 999. Accuracy will be measured as the percentage of correct subtractions.
Usual walk | 45-second
  fNIRS with walking trial 20m indoor course with 180-degree turns at each end and an instrumented gait mat in the middle.
Walk with the cognitive task (DT) | 45-second
  fNIRS with walking trial 20m indoor course with 180-degree turns at each end and an instrumented gait mat in the middle.

SECONDARY OUTCOMES:
Mobility - SPPB (Short Physical Performance Battery) | 9 months
  Evaluating participants' physical performance through a battery of tests including balance, walking speed, and chair stand tests.
Mobility - 4 m Gait Test | 9 months
  Measuring participants' gait speed over a 4-meter distance.
Mobility - Falls Efficacy Scale-International (FES-I) | 9 months
  Participants' fear of falling and confidence in performing daily activities without falling will be assessed using the Falls Efficacy Scale-International (FES-I).
  Scale: Scores range from 16 to 64, with higher scores indicating a greater fear of falling (worse outcome).
Mobility - Habitual Physical Activity and Real-World Gait | 9 months
  Monitoring participants' habitual physical activity and gait in real-world settings using an Axivity sensor taped to the lower back.
Mood- Geriatric Depression Scale (GDS | 9 months
  A 15-item questionnaire used to assess depressive symptoms in older adults. Scale: Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms (worse outcome).
Mood- SF-36 (Short Form Health Survey) | 9 months
  A 36-item questionnaire used to assess overall health-related quality of life, including emotional well-being.
  Scale: Scores range from 0 to 100, with higher scores indicating better health and well-being (better outcome).
anxiety- Geriatric Anxiety Inventory - Short Form (GAI-SF) | 9 months
  Questionnaire: Geriatric Anxiety Inventory - Short Form (GAI-SF). Scores range from 0 to 20, with higher scores indicating greater anxiety (worse outcome).
apathy | 9 months
  The Apathy Scale is used to assess the level of apathy in participants. Scale: Scores range from 0 to 42, with higher scores indicating greater apathy (worse outcome).
Functional Activity Questionnaire | 9 months
  Functional Activity Questionnaire- Scores range from 0 to 30, with higher scores indicating greater difficulty in performing daily activities (worse outcome).
Cognitive Function - Motor Screening Task | 9 months
  Assessment: The Motor Screening Task will evaluate participants' basic motor abilities using a computerized test. Scores range from 0 to 100, with higher scores indicating better motor function.
Cognitive Function - Reaction Time | 9 months
  Reaction Time will be measured to assess the speed of cognitive processing using a computerized test.
  Scale: Reaction time is measured in milliseconds, with lower times indicating faster cognitive processing (better outcome).
cognitive Function | 9 months
  battery to minimize procedural learning. ll tests have excellent psychometric properties and normative data suitable for our sample. validated battery of computerized tests (CANTAB Connect Research).Specific tests include the Motor Screening Task, Reaction Time, Paired Associates Learning, Spatial Working Memory, Pattern Recognition Memory, Delayed Matching to Sample, and Rapid Visual Information Processing. Additionally, participants will complete the MoCA, RAVLT, and Category and Phonemic Fluency tests.
Cognitive Function - Paired Associates Learning | 9 months
  The Paired Associates Learning test will evaluate memory function by assessing participants' ability to recall associations between objects and locations.
  Scale: Scores range from 0 to 100, with higher scores indicating better memory function.
Cognitive Function - Spatial Working Memory | 9 months
  Spatial Working Memory will be assessed using a computerized test to evaluate participants' ability to retain and manipulate spatial information.
  Scale: Scores range from 0 to 100, with higher scores indicating better working memory.
Cognitive Function - Pattern Recognition Memory | 9 months
  Pattern Recognition Memory will be tested to measure participants' visual memory and pattern recognition abilities.
  Scale: Scores range from 0 to 100, with higher scores indicating better pattern recognition. Scale: Scores range from 0 to 100, with higher scores indicating better working memory.
Cognitive Function - Delayed Matching to Sample | 9 months
  Delayed Matching to Sample will be used to evaluate visual memory and matching abilities after a delay.
  Scale: Scores range from 0 to 100, with higher scores indicating better matching abilities.
  Scale: Scores range from 0 to 100, with higher scores indicating better working memory.
Cognitive Function - Rapid Visual Information Processing | 9 months
  The Rapid Visual Information Processing task will assess sustained attention and visual processing speed.
  Scale: Accuracy is scored from 0 to 100, with higher scores indicating better sustained attention. Reaction time is measured in milliseconds, with lower times indicating faster processing. Scale: Scores range from 0 to 100, with higher scores indicating better working memory.
Cognitive Function - Montreal Cognitive Assessment (MoCA) | 9 months
  The MoCA will be used to evaluate global cognitive function across multiple domains.
  Scale: Scores range from 0 to 30, with higher scores indicating better cognitive function.
Cognitive Function - Rey Auditory Verbal Learning Test (RAVLT) | 9 months
  The RAVLT will assess verbal memory through recall and recognition tasks. Scale: Scores range from 0 to 15 for immediate recall, with higher scores indicating better memory performance. Scale: Scores range from 0 to 30, with higher scores indicating better cognitive function.
Cognitive Function - Category and Phonemic Fluency Tests | 9 months
  These tests will evaluate participants' semantic knowledge and word retrieval abilities.
  Scale: Scores represent the number of correct words generated within a time limit, with higher scores indicating better fluency. Scale: Scores range from 0 to 30, with higher scores indicating better cognitive function.
Height | 9 months
  Height will be measured in meters.
Weight | 9 months
  Weight will be measured in kilograms.
Medical History | 9 months
  Medical History
Blood Pressure | 9 months
  Blood Pressure

IPD SHARING:
Plan to Share IPD: No